CLINICAL TRIAL: NCT06519825
Title: The Effect of Inspiratory Muscle Strength Training on Posture, Respiratory Functions, Respiratory Muscle Strength and Performance in Healthy Adults With Forward Head Posture
Brief Title: The Effect of Inspiratory Muscle Strength Training in Healthy Adults With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, Lecturer, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024 - 41
Record Dates: First submitted 2024-07-02; First posted 2024-07-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-11

CONDITIONS: Posture
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Forward head posture-Study (Experimental): participants with a forward head posture who will undergo an exercise program
  Interventions: Other: Exercise
- Forward head posture-Control (No Intervention): participants with forward head posture who will not perform an exercise program
- Control group (No Intervention): control group without forward head posture

INTERVENTIONS:
Other: Exercise — Inspiratory muscle strength training program will be applied to the FHP-C group for 7 days/6 weeks.
  Arms: Forward head posture-Study

SUMMARY:
Forward head posture (FHP) is defined as the position in which the head is in front of the shoulder and is one of the most common musculoskeletal problems caused by the increasing use of computers and smartphones. Posture analysis, pulmonary function test, respiratory muscle strength and endurance assessment, and performance test will be performed as the initial evaluation for those who meet the inclusion criteria and volunteer to participate in the study. Participants with a craniovertebral angle of 50 degrees and less than 50 degrees will be included in the head forward posture (FHP, n=34) group, and participants with an angle of more than 50 degrees will be included in the control group (CG, n=34).Participants with HFP will be randomly divided into two groups as study (FHP-S, n=17) and control (FHP-C, n=17). An inspiratory muscle strength training program will be applied to the FHP-C group for 7 days/6 weeks. All assessments performed before the training will be repeated after 6 weeks of inspiratory muscle strength training. No inspiratory muscle strength training will be applied to the FHP-C group. Participants in the CG group will not undergo any additional assessment or training.

DETAILED DESCRIPTION:
Forward head posture (FHP) is defined as the position in which the head is in front of the shoulder and is one of the most common musculoskeletal problems caused by the increasing use of computers and smartphones. Posture analysis, pulmonary function test, respiratory muscle strength and endurance assessment, and performance test will be performed as the initial evaluation for those who meet the inclusion criteria and volunteer to participate in the study. Participants with a craniovertebral angle of 50 degrees and less than 50 degrees will be included in the head forward posture (FHP, n=34) group, and participants with an angle of more than 50 degrees will be included in the control group (CG, n=34).Participants with HFP will be randomly divided into two groups as study (FHP-S, n=17) and control (FHP-C, n=17). An inspiratory muscle strength training program will be applied to the FHP-C group for 7 days/6 weeks. All assessments performed before the training will be repeated after 6 weeks of inspiratory muscle strength training. No inspiratory muscle strength training will be applied to the FHP-C group. Participants in the CG group will not undergo any additional assessment or training.

ELIGIBILITY:
Inclusion Criteria:

* Cranio-vertebral angle (CVA) of 50 degrees and less than 50 degrees

Exclusion Criteria:

* Diagnosed respiratory, neurological, orthopedic, psychiatric or cardiac problems
* Have any infection at the time of assessment and training,
* Having any limitation that prevents assessment and training
* Pregnancy or breastfeeding
* Having a history of neck trauma
* Having undergone lumbar-neck surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Craniovertebral angle | Baseline
  Where a line drawn from the tragus of the ear to the C7 vertebra intersects a horizontal line, the CV angle is formed.
Sagittal head tilt | Baseline
  This angle, which is formed between a line from the canthus of the eye and the tragus of the ear and the horizontal, is a measure of the posture of the upper cervical spine.
Sagittal shoulder-C7 angle | Baseline
  Where a horizontal line passing through the lateral shoulder meets the line drawn from C7 to the lateral shoulder, the point of intersection forms the sagittal shoulder-C7 angle
Kyphosis angle measurement | Baseline
  The spinous processes of C7 and T12 vertebrae will be marked by a marker (reflector). Extensions of these reflectors will be taken and perpendicular lines will be drawn to these extensions. The angle formed by the intersection of the perpendicular lines will be measured as the thoracic kyphosis angle

SECONDARY OUTCOMES:
Pulmonary Function Tests- FEV1/FVC | Baseline
  Evaluation of FEV1/FVC ratio MicroQuark® computer-based USB spirometer will be used to assess the respiratory function of the participants. The person will be asked to take a few normal breaths followed by as deep a breath as possible and instructed to exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- FVC | Baseline
  Evaluation of Forced Vital Capacity (FVC) MicroQuark® computer-based USB spirometer will be used for FVC evaluation. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- FEV1 | Baseline
  Evaluation of Forced Expiratory Volume in 1 second (FEV1) MicroQuark® computer-based USB spirometer will be used for FEV1 evaluation. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- PEF | Baseline
  Evaluation of Peak Expiratory Flow (PEF) MicroQuark® computer-based USB spirometer will be used for PEF evaluation. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- MVV | Baseline
  Maximum voluntary ventilation (MVV) MicroQuark® computer-based USB spirometer will be used for MVV evaluation. Then the participant will take the disposable bacteria filter mouthpiece between his lips and holds it tightly. The person will be asked to deeply and rapidly breaths for 10 to 15 seconds.
Respiratory Muscle Strength | Baseline
  During the measurements, the nose of the individual participating in the study will be covered with a nose clip. During the maximal inspiratory pressure (MIP) measurement, the participants will be asked to inspire quickly and deeply with maximum effort after maximum expiration. For maximal expiratory pressure (MEP), the participant will be asked to expire quickly and deeply after maximum inspiration.
Sport performance | Baseline
  Subjects run back and forth on a 20 m course and must touch the 20 m line; at the same time a sound signal is emitted from a prerecorded tape. Frequency of the sound signals is increased 0.5 km h-1 each minute from a starting speed of 8.5 km h-1. When the subject can no longer follow the pace, the test is stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin A. Güzel, Prof. Dr., Study Director — Gazi University
Locations (1):
- Niğde Ömer Halisdemir Üniversitesi, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No